CLINICAL TRIAL: NCT00431340
Title: A Phase II Study of Belinostat in Combination With Bortezomib in Patients With Relapsed, Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to dose limiting toxicity
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PXD101-CLN-16
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; myeloma; plasma cell myeloma; bone marrow cancer; myelomatosis; Kahler's disease; PXD101; belinostat; bortezomib
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Bone Marrow Neoplasms | interventions — belinostat

INTERVENTIONS:
Drug: PXD101

SUMMARY:
This open-label study will assess anti-tumor activity and safety of belinostat in combination with bortezomib (Velcade®) in multiple myeloma patients refractory to or relapsed from at least one prior bortezomib-containing regimen. Subjects will be administered both PXD101 and bortezomib on the same days: i.e. days 1, 4, 8, and 11 of a 3-week cycle, for up to 8 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma.
* Status of refractory to or relapsed from at least one prior bortezomib-containing regimen.
* Progressive disease.
* Age >= 18 years.
* Karnofsky performance status >= 60%
* Acceptable liver function:

  * Bilirubin =< 1.5 x ULN (upper limit of normal)
  * Aspartate transaminase (AST) and alanine transaminase (ALT) =< 3 x ULN
* Acceptable hematologic status:

  * Absolute Neutrophil Count (ANC) >= 1.5 x 109/L
  * Platelet count >= 100 x 109/L
  * Hemoglobin >= 9 g/dL
  * Coagulation status PT-INR/PTT =< 1.5 x ULN or in the therapeutic range if on anticoagulation therapy. (PT-INR/PTT= prothrombin - international normalized ratio / prothrombin time)
  * Serum potassium within normal range.
* Estimated life expectancy greater than 3 months.
* Signed, written IRB (institutional Review Board)-approved informed consent.

Exclusion Criteria:

* Non-secretory multiple myeloma or symptomatic amyloidosis.
* Hypersensitivity to bortezomib, boron, or mannitol.
* Less than 4 weeks since prior chemotherapy, radiotherapy, endocrine therapy, or immunotherapy, except if disease is rapidly progressing.
* Less than 4 weeks since prior use of other investigational agents.
* Serious concomitant systemic disorders (e.g. active infection).
* Significant cardiovascular disease.
* Marked baseline prolongation of QT/QTc (corrected QT interval)interval.
* Central nervous system disorders requiring neuroleptics / anti-convulsants.
* Peripheral sensory neuropathy of ≥ Grade 2
* Renal insufficiency defined as a creatinine clearance of < 30 ml/min.
* Non-willingness to use effective contraceptive methods for patients of child-bearing age / potential.
* Pregnant or breast-feeding women.
* Known HIV positivity.
* Prior treatment with belinostat (PXD101), or any other HDAC (histone deacetylase) inhibitor.
* Altered mental status which precludes an understanding of the Informed Consent Document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Objective response rate of belinostat administered in combination with bortezomib in multiple myeloma subjects who are refractory to or have relapsed from at least one prior bortezomib-containing regimen.
Safety of belinostat plus bortezomib.

SECONDARY OUTCOMES:
Duration of response, time to response (TTR), and time to progression (TTP).
Effect on biomarkers of bone metabolism. Effect on disease-related bone pain.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Oncotherapeutics, West Hollywood, California
  - Center for cancer and blood disorders, Bethesda, Maryland
  - Baylor University Medical Center, Dallas, Texas